CLINICAL TRIAL: NCT03021200
Title: Use of Laser Fluorescence With Spy Elite, Pinpoint and Firefly Robotic Platform Systems in Cancer Surgical Treatment
Brief Title: Laser Fluorescence in Cancer Surgical Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Fundação Faculdade de Medicina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP953/16
Record Dates: First submitted 2017-01-04; First posted 2017-01-13 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Esophageal Cancer; Gastric Cancer; ColoRectal Cancer; Prostatic Neoplasms; Uterine Cancer; Head and Neck Cancer; Breast Neoplasm
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Uterine Neoplasms; Head and Neck Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Indocyanine green in Conventional Oncological Surgery (Experimental): Use of indocyanine green laser fluorescence angiography (AFLIICG) platforms (SPY-Elite) for conventional oncological surgeries
  Interventions: Device: Green indocianine
- Indocyanine green in minimally invasive Oncological Surgery (Experimental): Use of indocyanine green laser fluorescence angiography (AFLIICG) platforms (Pinpoint) for minimally invasive oncological surgeries
  Interventions: Device: Green indocianine
- Indocyanine green in robot-assisted Oncological Surgery (Experimental): Use of indocyanine green laser fluorescence angiography (AFLIICG) platforms (Firefly) for robot-assisted oncological surgeries
  Interventions: Device: Green indocianine

INTERVENTIONS:
Device: Green indocianine — Laser fluorescence using green indocianine guiding the surgical procedure.

SUMMARY:
The use of fluorescence for real-time evaluation of organ and tissue vascularization and lymph node anatomy is a recent technology with potential for the surgical treatment of cancer. The real-time analysis of tissue vascularization allows immediate identification to the surgeon of areas with greater or lesser blood circulation, favoring surgical decision making and prevention of complications related to tissue ischemia (necrosis, dehiscences and infections). It is a technology with potential application in the areas of Digestive Surgery, Repairing Plastic Surgery in Oncology, Head and Neck Surgery. In addition, fluorescence can be used as a method to identify lymph node structures of interest in the oncological treatment of patients with urologic, gynecological and digestive tumors.

Introduced by Pestana et al. In the late 2000s, the perfusion mapping system through intraoperative indocyanine assisted laser angiography (SPY Elite System © LifeCell Corp., Branchburg, N.J.) had its initial application in repairing surgery after breast cancer treatment. The method proved to be useful in the prevention of ischemic and infectious complications in cancer surgery. Pestana, in a prospective clinical series of 29 microsurgical flaps used in several reconstructions, observed a single case of partial loss of the flap, the present technology having a relevant role in intraoperative decision making. In the same year, Newman et al. The first application of the system in breast reconstruction surgery. In an initial series of 10 consecutive cases of reconstruction with microsurgical flaps, in 4 cases the system allowed the intraoperative identification of areas of low perfusion, thus changing the surgical procedure. According to the authors, there was a 95% correlation between indocyanine laser assisted and subsequent development of mastectomy skin necrosis, with sensitivity of 100% and specificity of 91%. Similarly, Murray et al. Evaluated the intraoperative perfusion, however, of the areola-papillary complex in patients submitted to subcutaneous mastectomies with satisfactory results in terms of predictability of cutaneous circulation. Other authors in larger clinical series and evaluating other procedures have observed valid results in terms of prevention of complications.

Vascular perfusion of anastomoses and fistulas following bowel surgery for cancer remain a serious and common complication. These fistulas can be caused by insufficient perfusion of the intestinal anastomosis. Intraoperative angiography with indocyanine assisted laser can be used to visualize the blood perfusion following intravenous injection of the indocyanine green contrast. Several groups reported the ability to assess blood perfusion of the anastomotic area after bowel surgery. Although they studied retrospectively, Kudszus and colleagues described a reduction in the risk of revision due to fistula in 60% of patients whose anastomosis was examined using laser fluorescence angiography compared to historically paired patients without this method. The same principle can be used to evaluate the tubulized stomach to be transposed to the cervical region after subtotal esophagectomy.

Currently, fluorescence-guided sentinel lymph node mapping has been studied in breast cancer as well as investigative character in colorectal cancer, skin cancer, cervical cancer, vulvar cancer, head and neck, lung cancer, penile cancer, cancer Endometrial cancer, gastric cancer and esophageal cancer.

These early studies demonstrated the feasibility of this methodology during surgery. Comparison of laser fluorescence images on blue dyes indicate that fluorescence images can replace blue dyes because they exceed them due to increased tissue penetration depth and absence of staining in the patient and cleaning of the operative field.

To date, there are no clinical studies involving intraoperative perfusion mapping and identification of lymph node structures with the SPY Elite System © system or other platforms (Pinpoint or Firefly) in Brazil that evaluate the Brazilian population. In an objective way the influence of this technology as predictive in the better or worse evolution of the oncologic surgery as well as in the prevention of the local ischemic complications by means of intraopeal change of conduct

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer and indication for one of the following surgeries:
* Low Anterior Resection
* Esophagectomy
* Lymphadenectomy
* Prostatectomy
* Pelvic or paraortic lymphadenectomy
* Surgery of head and neck with indication of supraclavicular flap
* Mastectomy followed by immediate or late breast reconstruction

Exclusion Criteria:

* Patients with a history of adverse reaction or known allergy to contrast, or iodine tinctures;
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2016-07-12 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
Intestinal Anastomosis Fistula | 3 years
  Intestinal Anastomosis Fistula Rate in oncologic resection of intestinal tumors
Esophageal fistula | 3 years
  Esophageal reconstruction fistula rate in esophagectomies
positive lymph nodes | 3 years
  The number of fluorescence-positive lymph nodes per patient
lymph nodes detected by pathology | 3 years
  The number of lymph nodes detected by pathology per patient
Mastectomy Skin Necrosis | 3 years
  Mastectomy Skin Necrosis Rate in Breast Reconstructions
Breast Implant Extrusion | 3 years
  Breast Implant Extrusion Rate in Breast Reconstructions
Surgical Site Infection in Breast Reconstructions | 3 years
  Surgical Site Infection Rate in Breast Reconstructions
Skin Necrosis in Head and Neck Reconstruction | 3 years
  Skin Necrosis Rate in Supraclavicular snip in Head and Neck Reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Ulysses Ribeiro, MD, Principal Investigator — Instituto do Cancer do Estado de Sao Paulo
Locations (1):
- Ulysses Ribeiro Junior, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No